CLINICAL TRIAL: NCT02960152
Title: Periodontal Impact of Eating Disorders (the PERIOED Study)
Acronym: PERIOED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Paris 7 - Denis Diderot (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Hélène Rangé, Dr, University Paris 7 - Denis Diderot
Other Study IDs: 13588
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Periodontal Diseases; Eating Disorder; Anorexia Nervosa; Bulimia Nervosa
Keywords: periodontitis
MeSH Terms: conditions — Periodontal Diseases; Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Anorexia Nervosa: interview and periodontal full-mouth examination
  Interventions: Other: diagnostic
- Bulimia Nervosa: interview and periodontal full-mouth examination
  Interventions: Other: diagnostic
- Control: interview and periodontal full-mouth examination
  Interventions: Other: diagnostic

INTERVENTIONS:
Other: diagnostic — full-mouth periodontal examination

SUMMARY:
This study evaluated the periodontal status of patients suffering from eating disorders (anorexia nervosa and bulimia nervosa). The work hypothesis is that eating disorder patients have a higher risk for periodontal diseases than non-eating disorder subjects.

DETAILED DESCRIPTION:
Eating disorders have been associated with poor oral health. However, the relationship between eating disorders and periodontal diseases is less-established. Participants will be periodontally assessed using a full-mouth clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* In and out eating disorder patients
* Subject with a diagnosis of anorexia nervosa or bulimia nervosa for at least 5 years
* Subject affiliated to the French social insurance

Exclusion Criteria:

* Subject who do not speak French
* Subject who is not able to read and/or understand the information form
* Subject who take anti-inflammatory medications or antibiotics at dental examination
* Subject who has received any dental treatment that could interfere with the periodontal status 3 month before the clinical examination (scaling and root planning, orthodontic treatment ongoing)
* Subject who has less than 10 teeth

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients suffering from eating disorders referred to the Psychiatric and Addiction department at the Paul Brousse Hospital (Villejuif, France)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Loss (CAL) | at examination day
  Periodontal probing depth and gingival recession are measured in millimeters using a manual periodontal probe (HuFriedy PCP UNC 15 probe, Chicago, IL, USA). At the clinical examination day, CAL is calculated as periodontal probing depth (mm) + gingival recession (mm) at 6 sites per tooth.

SECONDARY OUTCOMES:
gingival inflammation | at examination day
  Gingival inflammation is measured by bleeding on probing score (%) at 6 sites per tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bouchard, DDS, PhD, Study Chair — Paris Diderot University
Locations (2):
- France (2):
  - Rothschild Hospital, Paris
  - Paul Brousse Hospital, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available on request.